CLINICAL TRIAL: NCT01060358
Title: Neuromuscular Neutral Zones in Humans: A New Method to Assess Spinal Stability
Brief Title: Assessment of Spinal Stability
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 08-0063; 2586067 (Other: UC Denver Project Number); K99AT004983 (NIH)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2010-01

CONDITIONS: Spine Stability; Low Back Pain
Keywords: lumbar spine; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- healthy: Healthy and active men and women between 21 and 45 years old with no history of low back pain or low back injury.
  Interventions: Procedure: method (non-surgical) to measure neuromuscular neutral zones

INTERVENTIONS:
Procedure: method (non-surgical) to measure neuromuscular neutral zones

SUMMARY:
The purpose of this study is to verify the existence of neuromuscular neutral zones(NNZs) in humans, and develop non-invasive techniques to measure intervertebral kinematics of the lumbar spine. The results will be used to accurately quantify NNZs in humans, and provide a foundation for clinical trials on low back pain patients using this methodology.

ELIGIBILITY:
Inclusion Criteria:

* 21-45 years of age - typical working age in physically demanding jobs
* no history of low back injury or musculoskeletal disorder in the past one year
* any activity history: sedentary, active, or non-athletic, and 4) any ethnic background or race
* body mass index score less than 30

Exclusion Criteria:

* Younger than 21 or older than 45 years old (range not relevant to majority of physical labor force)
* previous injury, disorder, or illness related to the low back
* professional athletes
* professional workers engaged in physical labor (e.g., roofers, loaders/unloaders in warehouses, tile/concrete layers, etc.)
* pregnancy

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healty men and women between 21 and 45 years old with no history of low back pain of low back injury.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
neuromuscular neutral zones | one year

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Davidson, Ph.D., Principal Investigator — University of Colorado, Denver; Moshe Solomonow, Ph.D., M.D. (hon), Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States